CLINICAL TRIAL: NCT06035549
Title: Development of a Culturally Tailored Digital Resilience-Building Intervention for East Asian Immigrants With Cancer to Facilitate Advance Care Planning Discussions
Brief Title: Resilience in East Asian Immigrants for Advance Care Planning Discussions
Status: Recruiting | Type: Observational
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Rockefeller University (Other)
Responsible Party: Principal Investigator, Li-Ting Longcoy, Postdoctoral Research Associate/Principal Investigator, University of Illinois at Chicago
Other Study IDs: 2023-0560; KC_Awd_114452 (Other: University of Illinois at Chicago)
Record Dates: First submitted 2023-09-06; First posted 2023-09-13 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Neoplasms; Advance Care Planning
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Culturally Tailored Digital Resilience-Building: The culturally tailored resilience-building materials will be provided to East Asian immigrants with cancer and their family caregivers.
  Interventions: Behavioral: Culturally Tailored Digital Resilience-Building
- Religious leaders: Religious leaders providing spiritual care to Asian Americans
  Interventions: Behavioral: Semi-structured interviews

INTERVENTIONS:
Behavioral: Culturally Tailored Digital Resilience-Building — The Culturally Tailored Digital Resilience-Building materials include an introduction to advance care planning and resilience skills that specifically address cultural beliefs and barriers.
  Groups: Culturally Tailored Digital Resilience-Building
Behavioral: Semi-structured interviews — Semi-structured interviews with religious leaders who provide spiritual care to Asian Americans/immigrants.
  Groups: Religious leaders

SUMMARY:
The purpose of the study is to develop a culturally tailored digital resilience-building intervention to help East Asian immigrants engage in advance care planning discussions with their family caregivers.

DETAILED DESCRIPTION:
Advance care planning (ACP) is a process to facilitate decision-making for future care and document values and preferences. However, the advance directive completion rates in East Asian Americans are low, which may extend to disparities in end-of-life care, including rates of hospice use and prevalence of unwanted aggressive treatments. To address this, this study uses information technology to develop a culturally tailored digital resilience-building intervention with and for East Asian immigrants to help them engage in ACP discussions. There are two aims of this study: (1) Conduct semi-structured interviews with a total of 30 religious leaders to identify the barriers and facilitators associated with discussing ACP and death-related topics with immigrants from China/Taiwan, Japan, and Korea and (2) Develop a culturally tailored digital resilience-building intervention using think-aloud interviews with 27 pairs of East Asian immigrants with cancer and their family caregivers (9 pairs each for immigrants from China/Taiwan, Japan, and Korea).

ELIGIBILITY:
Inclusion Criteria for Religious Leaders:

* Age ≥ 18 years
* Serving as a chaplain or religious leader at a healthcare setting or religious organization
* Having experience providing pastoral or spiritual care to Chinese, Japanese, and Korean Americans in the US
* Being able to read and respond to questions in English, Mandarin, Cantonese, Japanese, or Korean.

Exclusion criteria: Not willing to provide consent.

Inclusion Criteria for Patients:

* Age ≥ 18 years
* Having a cancer diagnosis
* Likely self-identifying as a Chinese, Japanese, or Korean American/immigrant
* Being able to read and respond to questions in either English, Mandarin, Japanese, Korean, or Chinese dialects, such as Cantonese, Shanghai, Taishanese, or Taiwanese.

Exclusion Criteria for Patients:

* Having cognitive impairment per the Short Portable Mental Status Questionnaire with more than three errors

Inclusion Criteria for Family Caregivers:

* Age ≥ 18 years
* Being able to read and respond to questions in either English, Mandarin, Japanese, Korean, or Chinese dialects, such as Cantonese, Shanghai, Taishanese, or Taiwanese
* Having a family member who is likely to self-identify as a Chinese, Japanese, or Korean American/immigrant and has been diagnosed with cancer

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Religious leaders providing spiritual care to Asian Americans/immigrants or Asian Americans/immigrants living with cancer
Sampling Method: Non-Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2023-10-27 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Usability | Immediately at the end of the think-aloud interview
  Use the System Usability Scale (range: 0-100) to assess the usability of the intervention. Higher scores indicate greater perceived usability by users.

SECONDARY OUTCOMES:
Acceptability | Immediately at the end of the think-aloud interview
  Use the Acceptability E-scale to assess the acceptability of the intervention. Scale total scores range from 6 to 30, and higher scores indicate greater acceptance for the proposed intervention.

OTHER OUTCOMES:
Religious leaders experience | Immediately at the end of the interview
  An in-depth understanding of religious leaders' perspectives on barriers and facilitators to discussing death-related topics with immigrants from East Asia.

CONTACTS AND LOCATIONS:
Overall Officials: Li-Ting H. Longcoy, Principal Investigator — University of Illinois Chicago College of Nursing
Locations (1):
- University of Illinois Chicago, Chicago, Illinois, United States